CLINICAL TRIAL: NCT06112925
Title: Impact of Medication Therapy Management Intervention on Treatment Outcomes and Medication Adherence Among Adult Patients Comorbid With Diabetes Mellitus and Hypertension at Outpatient Clinics in Southwest Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: Impact of Medication Therapy Management Intervention on Treatment Outcomes and Medication Adherence Among Adult Patients Comorbid With Diabetes Mellitus and Hypertension at Outpatient Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mattu University (Other)
Responsible Party: Principal Investigator, Tadesse Sheleme Achalu, Lecturer, Mattu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MattuU
Record Dates: First submitted 2023-10-05; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Treatment outcomes; Medication adherence; Diabetes Mellitus and Hypertension; Southwest Ethiopia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Medication Adherence | interventions — Medication Therapy Management

STUDY DESIGN:
Intervention Model Description: There were two groups of study population.
Who Masked: Participant, Care Provider
Masking Description: The study participants and attending healthcare providers were blinded of participants' treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Therapy Management (Experimental): The patients attending hospitals assigned to interventional group received medication therapy management services in addition to usual care. The medication therapy management services was provided by the clinical pharmacists. The study participants and attending healthcare providers were blinded of participants' treatment group. The intervention was done at initial visit and repeated at 3rd and 6th month of the initial visit.
  Interventions: Other: Medication Therapy Management
- No Medication Therapy Management (No Intervention): The patients attending hospitals assigned to controlled group received usual care only. The usual care is patients' discussion with the attending physician, and nurse regarding their disease, medications, and subsequent appointments which may take approximately 5 minutes. Two consecutive follow-up visits were scheduled for 3rd month and 6th of initial visit for each patients in similar to interventional group.

INTERVENTIONS:
Other: Medication Therapy Management — The medication therapy management intervention was delivered via the five (5) core components which include medication therapy review, personal medication record, medication-related action plan, intervention, and documentation and follow-up. The interventions was also given via educating patients about diabetes, hypertension, complications of diabetes and hypertension, impact of having diabetes and hypertension, antidiabetes and antihypertensive medications, goals of therapy for diabetes and hypertension, health promoting behaviours (healthy diet, regular exercise, salt reduction, & smoking cessation), drug adherence, and self-monitoring of the diseases.
  Arms: Medication Therapy Management

SUMMARY:
The goal of this interventional study was to assess the impact of medication therapy management on treatment outcomes and medication adherence among adult patients comorbid with diabetes mellitus and hypertension at outpatient clinics in Southwest Ethiopia. The patients attending hospitals assigned to interventional group received medication therapy management services in addition to usual care.

DETAILED DESCRIPTION:
This study aimed to assess the impact of medication therapy management intervention on treatment outcomes and medication adherence among patients comorbid with diabetes mellitus and hypertension at outpatient clinics in Southwest Ethiopia. A cluster randomized controlled trial was conducted at outpatient clinics of public hospitals in Southwest Ethiopia from March to December, 2022. Hospitals were randomly assigned to either the interventional or the control group. The patients attending hospitals assigned to interventional group received medication therapy management services in addition to usual care and those attended hospital assigned to control group received the usual care only. A systematic random sampling technique was used to select the study participants from each hospital. The differences in proportion between the groups was determined using the Pearson chi-square. The independent sample t-test was be done to compare means between groups and paired t-test was used to compare means in between intervention and controlled group. The p-value of < 0.05 was used as a cut-off point to declare statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* age is greater than or equal to 18 years
* diagnosed with both diabetes mellitus and hypertension

Exclusion Criteria:

* unwillingness to participate
* mentally disabled
* lost to follow-up
* change follow up site
* pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in percentage of of glycemic control, blood pressure control and medication adherence among adult patients comorbid with diabetes mellitus and hypertension at outpatient clinics in Southwest Ethiopia | It was a 6 months study period
  The proportion of patients who achieved good glycemic control changed from 15.5% to 43.3% from baseline to the end of the study in the intervention group. The current study also observed that the percentage of intervention group participants at the goal increased from 36.6% to 60.3% from baseline to 6-month.The adherence rate in the intervention group increased by 50% while remaining fairly constant in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Mattu Univesity, Addis Ababa, Mettu, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Analysis done in group, not in individual. So, individual data will not be shared.